CLINICAL TRIAL: NCT05425277
Title: Assessing the Effectiveness of a Low-Cost, Evidence-Based Naturalistic Developmental Behavioral Intervention (NDBI) in IDEA Part C Early Intervention Settings
Brief Title: Assessing the Effectiveness of Reciprocal Imitation Teaching in Part C Early Intervention Settings (Sprout Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wendy Stone, Professor, College of Arts & Sciences: Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007803; W81XWH1910293 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2022-06-12; First posted 2022-06-21 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIT Training Group (Experimental): Providers in the RIT group (n=30) will receive an 8-hour virtual workshop (2 half-days) on RIT implementation and caregiver coaching. Each provider will invite 2 families in their caseload to participate in the study. Providers will coach families in the use of RIT. One intervention session for each enrolled family will be videotaped and scored for RIT fidelity.
  Interventions: Behavioral: Reciprocal Intervention Teaching (RIT)
- Daily Routines (Active Comparator): Providers in the Routines Control group (n=30) will receive a 3-hour virtual workshop focused on helping providers coach caregivers on how to increase children's participation and social engagement during everyday home routines (i.e., snack time, bedtime, bath time, and family playtime). Each provider will invite 2 families in their caseload to participate in the study. One intervention session for each enrolled family will be videotaped and scored for RIT fidelity to ensure contamination has not occurred and the control condition providers are not utilizing RIT strategies.
  Interventions: Behavioral: Daily Routines

INTERVENTIONS:
Behavioral: Reciprocal Intervention Teaching (RIT) — RIT is a relatively straightforward, brief NDBI. It employs four simple strategies to target motor imitation and initiating joint attention during play: (1) contingent imitation of the child's verbal and nonverbal behavior, (2) linguistic mapping, (3) direct elicitation of object and gesture imitation following the child's interest, and (4) contingent reinforcement. It has been used at low intensities (e.g., 1-3 hours per week) over short periods of time (e.g., 10-12 weeks) to produce robust changes in pivotal social-communicative skills. RIT is easy to learn and can be implemented with fidelity by undergraduate-level therapists with limited backgrounds in ASD, as well as by caregivers and siblings.
  Arms: RIT Training Group
Behavioral: Daily Routines — The Routines webinar was adapted from a web-based tutorial developed by PI Stone and colleagues (Ibanez et al., 2018). The webinar covers topics such as why everyday routines are important, especially for children with ASD, specific steps for increasing children's participation in routines, and how to use strategies such as visual supports to clarify expectations, and provides numerous video examples of caregivers using different strategies. Providers are also given access to a video library of caregivers using the Daily Routines strategies with their children, as well as a workbook to use with families during treatment.
  Arms: Daily Routines

SUMMARY:
Despite strong consensus that early, specialized intervention for children with Autism Spectrum Disorder (ASD) can have a dramatic impact on outcomes, the public health system's capacity to provide such services is severely challenged by the rapid rise in ASD prevalence. The goal of this research project is to improve services and outcomes for children with early signs of ASD by testing the effectiveness of a brief, inexpensive training on EI providers' ability to deliver an evidence-based, caregiver-mediated intervention that can improve providers' comfort and effectiveness in working with families of children with social communication concerns, as well as improving child and family outcomes.

DETAILED DESCRIPTION:
Despite strong consensus that early, specialized intervention for children with Autism Spectrum Disorder (ASD) can have a dramatic impact on outcomes, the public health system's capacity to provide such services is severely challenged by the rapid rise in ASD prevalence. The long-term goal of this study is to improve services and outcomes for children with early signs of ASD by testing the effectiveness of training EI providers to deliver an evidence-based, inexpensive, caregiver-mediated intervention that can improve child and family outcomes as well as mitigate the substantial economic costs associated with ASD. This research will take place within an existing community-based infrastructure: the Part C Early Intervention (EI) service delivery system. Part C is publicly funded, available throughout the country, and serves children under age 3 who have developmental delays or disabilities, and their families. Currently, the effectiveness of EI services is limited by high practice variation and infrequent use of evidence-based interventions. The study objective is to improve services and outcomes for children with early signs of ASD and their families. Toward that end, the investigators are conducting a randomized controlled trial (RCT) examining the effectiveness of training EI providers to deliver Reciprocal Imitation Training (RIT), as compared to an active control condition. RIT is a naturalistic developmental behavioral intervention (NDBI) that is ideally suited for EI settings because it is low intensity, play-based, easy to learn and implement, and can be taught to families for their independent use, thus increasing intervention dosage. The investigators will conduct this study within the context of an effectiveness-implementation hybrid type 1 design to gather evidence that will be essential for implementing RIT in other communities if it is found to improve child and caregiver outcomes.

EI providers will be randomly assigned to either the RIT training (n=30) or an active control condition (n=30). Providers in both conditions will complete surveys about their caseloads and intervention practices at 5 time points, once before their training workshops and four times after the workshop (1, 3, 6, and 12 months post-training). Providers assigned to the RIT training condition will receive an 8-hour virtual workshop on the rationale for, and implementation of, RIT with families, with an emphasis on caregiver coaching. Providers assigned to the active control condition ('Daily Routines') will receive a 3-hour virtual workshop on methods for helping caregivers increase their children's participation and social engagement during everyday home routines. Providers in this condition will be able to receive RIT training at the end of the study.

Providers in both conditions will also invite 2 families from their caseload to participate in this study. Caregiver recruitment and data collection will begin immediately after the training workshops are conducted with providers. Enrolled families must speak and read English or Spanish and have a child between 18 and 30 months for whom ASD is either suspected or confirmed. Caregiver participation involves having one EI session videotaped, completing survey measures at 3 time points, and conducting a play-based assessment in their homes (with coaching) at the same 3 time points: baseline, 3 months later, and 6 months post-baseline. The play-based assessment will measure children's motor imitation, social communication, caregiver fidelity to RIT, and caregiver use of child-centered interaction strategies. At the same 3 timepoints, caregivers will complete measures about their parenting stress and parenting self-efficacy, their child's social communication and language, and any additional services the child is receiving. The child's adaptive behavior will be measured via caregiver-interview at baseline and 6-months. Caregivers will also report on the 'top concerns' they have about their child at baseline, and will rate the severity of these concerns monthly thereafter. Family-level "RIT dosage" will also be measured via a weekly Dosage Log sent to caregivers via text message. Caregiver-reported satisfaction with treatment and the study, as well as caregiver-reported child ASD symptomatology will be collected at their final visit (6-months after enrollment).

ELIGIBILITY:
Inclusion Criteria:

EI Providers:

* Speak and read English
* Work at a participating Part C practice or agency
* Have an active caseload that includes at least two children with ASD or suspected ASD
* Are willing to invite families to participate in this study

Caregivers and Toddlers (recruited from EI provider caseloads):

* Caregivers speak and read English or Spanish
* Caregivers are at least 18 years of age
* Caregivers are willing and able to participate in intervention sessions and research tele-visits that are video-recorded by research staff
* Child receives services from one of the participating agencies and attends regular sessions with the enrolled provider
* Child is between 18 and 30 months of age at study entry
* Child has a diagnosis of ASD or displays social communication impairments consistent with ASD

Exclusion Criteria:

• Child has no severe visual, auditory, or physical impairments and no serious medical, genetic, or neurological conditions that would impede their ability to engage in RIT.

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Child Social Communication - In Vivo | Change from baseline to 6-month follow-up
  Change in in-vivo observation of child social communication will be assessed using the scored social communication items on the TELE-ASD-PEDS (TAP; Corona et al., 2021). There are 5 social communication items that can be scored 1-3 (range 5-15, with lower scores indicating better outcome).
Child Social Communication - Parent Report | Change from baseline to 6-month follow-up
  Change in parent reported child social communication will be assessed using three subscales from the the Parent Interview for Autism-Clinical Version (PIA-CV; Stone et al., 2003).The subscales that will be examined are: Social Relating (17 questions), Language Understanding (7 questions), and Nonverbal Communication (13 questions). These items can be scored 1-5 (range 37-185, with higher scores indicating better outcome).
Child Social Communication - Behaviorally Coded | Change from baseline to 6-month follow-up
  Change in behaviorally coded child social communication will be assessed using the observationally coded Weighted Frequency of Intentional Communication during a parent-child free play task (Yoder et al., 2009).
Child Motor Imitation - In Vivo | Change from baseline to 6-month follow-up
  Change in behaviorally observed motor imitation will be assessed using an adapted version of the Motor Imitation Scale (MIS; Stone et al., 1997). Five items with three trials each will be presented to the child. If a child receives a maximum score, the item is discontinued. Each trial can be scored 0-2 (range 0-10, with higher scores indicating better outcome).
Child Motor Imitation - Parent Report | Change from baseline to 6-month follow-up
  Change in parent reported motor imitation will be assessed using the Parent Interview for Autism-Clinical Version (PIA-CV; Stone et al., 2003). The Imitation subscale (4 items) will be examined. These items can be scored 1-5 (range 4-20, with higher scores indicating better outcome).
Provider Coaching of Caregivers in RIT Strategies | Change from baseline to 12-month follow-up
  Change in providers' use of caregiver coaching strategies will be assessed via provider self-report survey.
Caregiver Use of RIT Strategies | Change from baseline to 6-month follow-up
  Change in caregiver use of RIT strategies will be assessed via a caregiver-child activity in which caregivers are instructed to demonstrate the skills they learned from their (enrolled) EI provider; scoring will employ the RIT Fidelity Checklist (range 6-30, with higher scores indicating higher fidelity to RIT).

SECONDARY OUTCOMES:
Child Adaptive Behavior | Change from baseline to 6-month follow-up
  Change in child adaptive behavior will be assessed using the Vineland Adaptive Behavior Scale - Third Edition (Vineland-3; Sparrow et al., 2016). The Vineland-3 provides norm-referenced scaled scores for 11 skill areas (M = 10; SD = 3) as well as standard scores (M =100, SD = 15) for three adaptive domains, with higher scores indicating better outcome.
Child Language | Change from baseline to 6-month follow-up
  Change in child language will be assessed using the MacArthur Bates Communicative Development Inventory (MCDI; Fenson et al., 2007). The MB-CDI is scored from 0 to 100 percentile, with a higher percentile indicating better outcome.
Parenting Self-Efficacy | Change from baseline to 6-month follow-up
  Change in parenting self-efficacy will be measured using the Parenting Efficacy Scale (PES; Teti & Gelfand, 1991). The PES contains 10 items scored 1-4 (range 10-40, with higher scores indicating better outcome).
Parenting Stress | Change from baseline to 6-month follow-up
  Change in parenting stress will be measured using the Parenting Stress Index-Short Form (PSI-SF; Abidin, 1990). The PSI-SF contains 36 items scored 0-4 and total score is presented as a percentile (range 0-100 with lower scores indicating better outcome).
Caregiver Top Concerns | Change from baseline to 6-month follow-up
  Change in severity ratings of each individual caregiver's top concerns about their child will be measured using an adapted version of the Caregiver Top Problems assessment (TPA; Weisz et al., 2013). The three items are rated from 0-4 (range 0-12, with lower scores indicating better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Stone, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No